CLINICAL TRIAL: NCT05857345
Title: Assessing Gene Expression in Lactocytes Using Human Breast Milk as a Non-Invasive Source: A Pilot Study
Brief Title: Breastmilk as a Source of Lactocytes
Status: Completed | Type: Observational
Sponsor: University of Hohenheim (Other)
Responsible Party: Sponsor
Other Study IDs: Breastmilk
Record Dates: First submitted 2023-04-21; First posted 2023-05-12 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Breastmilk Collection; Micronutrients
MeSH Terms: conditions — Breast Milk Expression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lactating individuals: Lactating adults (age >= 18) with children aged 2 weeks to 6 month
  Interventions: Other: Collection of breastmilk

INTERVENTIONS:
Other: Collection of breastmilk — Collection of breastmilk and other information about the participant

SUMMARY:
The objective of this study is to determine the suitability of lactocytes derived from human breast milk for gene expression analysis, and to explore whether there are any correlations between gene expression and the micronutrient composition of breast milk.

DETAILED DESCRIPTION:
Participants will be included in the study if they are willing to express milk and if their child is between 2 weeks and 6 months old. Participants' feeding practices (exclusive breastfeeding/non-exclusive breastfeeding) and micronutrient supplementation will be recorded. On the day of donation, child's age, the health status of both the mother and child (sick/not sick), the time of sample collection, and the number of feeding sessions that have taken place since midnight will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to express breastmilk
* Breastfed infant aged between 2 weeks and 6 months

Exclusion Criteria:

* Not willing to express breastmilk
* Infant older or younger than specified

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Yes
Study Population: Lactating mothers in Germany
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2023-04-28 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2023-10-23 (Actual)

PRIMARY OUTCOMES:
Gene Expression | 6 month after completion
  Gene expression of cellular markers from various cell populations in breast milk, as well as expression of proteins involved in micronutrient transport will be investigated. Additionally, these gene expression patterns will be investigated over time.
Micronutrient Content | 6 month after completion
  Micronutrient content of breastmilk will be analyzed and whether changes occur over time

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hohenheim, Stuttgart, Germany

IPD SHARING:
Plan to Share IPD: No